CLINICAL TRIAL: NCT06084598
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Intravenously Administered BMS-986446 in Healthy Participants Including Healthy Participants of Japanese Ethnicity
Brief Title: A Study to Evaluate the Safety, Tolerability and Drug Levels of BMS-986446 in Healthy Participants and Healthy Participants of Japanese Ethnicity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN008-0016
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetics; Healthy Participants; Healthy Japanese Participants; BMS-986446; PRX005

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986446 (Experimental)
  Interventions: Drug: BMS-986446
- Placebo (Experimental)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986446 — Specified dose on specified days
  Arms: BMS-986446
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and drug levels of BMS-986446 in healthy participants including healthy participants of Japanese ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be of Japanese ethnicity (both biological parents are ethnically Japanese) for Part 1 and Part 2, Panel 2. No limitations on ethnicity apply to Part 2, Panel 1
* Participant is healthy, without any significant abnormalities in medical history, physical examination, ECGs, or clinical laboratory assessments determinations, as assessed by the investigator
* Body mass index (BMI) of at least 18 kg/m^2 but no more than 32 kg/m^2 at screening
* Body weight between 45 kg and 110 kg

Exclusion Criteria:

* Any clinically significant deviation from normal, as judged by the investigator
* Any major surgery within 90 days of study drug administration
* Participation in another interventional clinical trial concurrent with this study

Note: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to Day 85
Number of participants with vital sign abnormalities | Up to Day 85
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 85
Number of participants with physical examination abnormalities | Up to Day 85
Number of participants with body weight abnormalities | Up to Day 85
Number of participants with clinical laboratory abnormalities | Up to Day 85

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 85
Time of maximum observed plasma concentration (Tmax) | Up to Day 85
Area under concentration time curve from time 0 to time of last quantifiable concentration [AUC(0-T)] | Up to Day 85
Number of participants with anti-drug antibody (ADA) | Up to Day 85
Geometric mean ratios of Cmax | Up to Day 85
Geometric mean ratios of [AUC(0-T)] | Up to Day 85
Geometric mean ratios of area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT06084598.html